CLINICAL TRIAL: NCT01997398
Title: DBS Under General Anesthesia Without Neurophysiology: Initial Experience and Comparison To The Standard Technique
Brief Title: DBS Under General Anesthesia: Comparison To The Standard Technique
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Other Study IDs: 12BN123
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson's Disease
Keywords: Deep brain stimulation surgery under general anesthesia; Deep brain stimulation target accuracy; Deep brain stimulation for Parkinsons's disease; Deep brain stimulation functional outcomes; Deep brain stimulation quality of life outcomes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a growing trend in functional neurosurgery toward direct anatomical targeting for deep brain stimulation (DBS). This study describes a method and reports the initial experience placing DBS electrodes under general anesthesia without the use of microelectrode recordings (MER), using a portable head CT scanner to verify accuracy intra-operatively.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an established therapy for Parkinson's disease and tremor. The therapy was first introduced in the late 1980s, and was FDA approved in 1997. Over 100,000 patients have been treated with DBS, and the benefits have been confirmed through multicenter randomized controlled trials.

Traditional DBS is performed with the patient awake. Parkinson's patients are required to be off their Parkinson's medicine during awake DBS, and single-unit cellular recordings are performed to map the intended target. Electrophysiological mapping can require multiple brain penetrations. The surgery can last 4-6 hours. The surgeon uses a local anesthetic to numb the tissue where the incision is made, and mild sedatives are administered to ward off anxiety. The prospect of being awake on the operating table for brain surgery concerns some patients, as does the requirement to be off medicine.

There is growing interest in performing DBS under general anesthesia, whereby targets are selected anatomically (i.e., on MRI) rather than physiologically . So-called "asleep DBS" is performed with the patient under general anesthesia, and uses intraoperative CT imaging both to target and to verify accurate placement of DBS electrodes at the time of surgery. Asleep DBS eliminates the need for the patient to be kept awake and off medicine. The goal of Asleep DBS is to accurately place the electrodes at the target selected by the surgeon preoperatively, and this goal is accomplished through intraoperative imaging. Electrophysiological mapping is not performed.

The Asleep DBS program at Barrow Neurological Institute / SJHMC started in March 2012; the second institution world-wide to adopt the asleep technique developed by Dr. Kim Burchiel. Other institutions have performed asleep DBS within an MRI magnet to visualize the placement of the electrode. The "Burchiel technique" relies upon MRI-CT fusion algorithms to superimpose the leads, seen on CT, on the MRI which was used for planning.

While asleep DBS improves the patient experience, it is incumbent upon us to demonstrate that the functional outcomes are equivalent to those reported for traditional "awake" DBS. Further, despite common use of MRI-CT fusion, which is available on our neuronavigation systems, the evidence supporting this modality comes from the 1990s, primarily from Gamma Knife literature.

This study will include functional outcomes using established metrics for Parkinson's, capturing both motor function (Unified Parkinson's Disease Rating Scale) and quality of life (Parkinson's Disease Questionnaire-39). In addition, follow-up MRI imaging will allow us to verify that the true position of the DBS leads matches where we thought the leads were based on the intraoperative CT scan that was fused to the preoperative MRI. In other words, there is an error in placement that we see at the time of surgery (if we our inaccuracy is over 2 mm, we reposition the DBS lead). There is also an inherent inaccuracy with CT-MRI fusion. If these inaccuracies are compounded such that where we think we are at the time of surgery is far from where we actually are (as seen on the follow-up MRI of the brain), then CT-MRI fusion is not reliable and should not be used to verify lead placement.

ELIGIBILITY:
Inclusion Criteria:

* Patient's who have undergone DBS surgery under general anesthesia without electrophysiology, utilizing a portable head CT scanner to verify accuracy intra-operatively.

Exclusion Criteria:

* Patient's who have undergone DBS surgery awake, without general anesthesia and with electrophysiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected by CPT codes corresponding to bilateral DBS electrode placement placed under general anesthesia with Leksell sterotactic navigation, portable CT and without the use of microelectrode recordings (MER).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — BARROW NEUROLOGICAL INSTITUTE / SJHMC
Locations (1):
- St. Joseph's Hospiatl & Medical Center / Barrow Neurological Institute, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All consecutive Parkinson's disease (PD) patients undergoing bilateral GPi deep brain stimulation surgery (DBS) under general anesthesia from May, 2012 - November of 2013.
Pre-assignment Details: Patients with advanced Parkinson's disease eligible for deep brain stimulation (DBS) surgery
Groups:
- Bilateral GPi DBS Surgery Under General Anesthesia: Patients underwent bilateral Gpi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
Period: Overall Study
Arm/Group | Bilateral GPi DBS Surgery Under General Anesthesia
Started | 35
Completed | 34 (One patient took PD meds 3 hours prior to 6 mo. UPDRS testing and was excluded from the analysis.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Patients who underwent bilateral GPi DBS surgery under general anesthesia
Groups:
- DBS Under General Anesthesia: Patients with advanced Parkinson's disease who underwent bilateral globus pallidus interna (GPi) deep brain stimulation surgery under general anesthesia without the use of microelectrode recordings or intraoperative stimulation.
Arm/Group | DBS Under General Anesthesia
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11
Average duration of Parkinson's disease [Mean (Standard Deviation); unit: years] | 10.7 (10)

OUTCOME MEASURES:

1. Primary Outcome: "Off" and "On" Medication Unified Parkinson's Disease Rating III Score (UPDRS)
Description: A movement disorders clinician who had completed the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) training performed prospective baseline and 6-month postoperative assessments of motor function using the MDS modified UPDRS III on patients during both off-medication (PD medications held for 12 h) and on-medication states.
  UPDRS III motor scores range from 0 (no motor function deficit) to 132 (highest motor function deficit). There were no subscales.
Time Frame: pre-operatively and 6 months post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-DBS Bilateral GPi DBS Under General Anesthesia "Off" Med: "Off " medication UPDRS III scores of patients scheduled for bilateral Gpi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
  Off medication .
- Post-DBS Bilateral GPi DBS Under General Anesthesia "Off" Med: "Off" medication UPDRS III scores of patients who underwent bilateral Gpi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
- Pre-DBS Bilateral GPi DBS Under General Anesthesia "On" Med: "On" medication scores of patients scheduled for bilateral GPi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
- Post-DBS Bilateral GPi DBS Under General Anesthesia "On" Med: "On" medication scores of patients who underwent bilateral GPi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
Arm/Group | Pre-DBS Bilateral GPi DBS Under General Anesthesia "Off" Med | Post-DBS Bilateral GPi DBS Under General Anesthesia "Off" Med | Pre-DBS Bilateral GPi DBS Under General Anesthesia "On" Med | Post-DBS Bilateral GPi DBS Under General Anesthesia "On" Med
Number analyzed (Participants) | 35 | 34 | 35 | 34
units on a scale | 48.4 (13.8) | 28.9 (12.5) | 23.52 (10.4) | 22.56 (12.8)
Statistical Analysis 1: Comparison: Pre-DBS Bilateral GPi DBS Under General Anesthesia "Off" Med vs Post-DBS Bilateral GPi DBS Under General Anesthesia "Off" Med; Test type: Superiority or Other; p < 0.001, Repeated measures general linear models — Differences in baseline and 6-month postoperative scores were assessed using a series of repeated measures general linear models with a single within-subjects factor and no between-subjects factors

2. Secondary Outcome: Parkinson's Disease Quality-39 Score (PDQ-39)
Description: Effects on PDQ-39 scores 6 months following asleep DBS surgery as compared to pre-operative scores. Data from the PDQ-39 can be presented either subset scores or as a single total score. PDQ-39 measures patient quality of life indicators including mobility, activities of daily living, emotional well being, stigma, communication and bodily discomfort. Data from the PDQ-39 can be presented in either subset scores or as a single total score. The full range of the total PDQ-39 scores is from 0 ( no patient related symptoms, or quality of life unaffected) to 156 ( relates having symptoms ", or low quality of life).
  The subset score ranges are as follows:
  mobility: 0 (no patient related symptoms) to 40 (highest patient related symptoms). activities of daily living: 0 to 24; emotional well being: 0-24; stigma: 0-16; cognition: 0-16; communication: 0-12; bodily discomfort: 0-12.
Time Frame: pre-operatively and 6 months post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-DBS Bilateral GPi DBS Surgery Under General Anesthesia: Patients scheduled for bilateral Gpi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
- Post - DBS Bilateral GPi DBS Surgery Under General Anesthesia: Patients who underwent bilateral Gpi DBS surgery under general anesthesia using intraoperative computed tomography to assess lead placement accuracy.
Arm/Group | Pre-DBS Bilateral GPi DBS Surgery Under General Anesthesia | Post - DBS Bilateral GPi DBS Surgery Under General Anesthesia
Number analyzed (Participants) | 35 | 34
units on a scale | 50.3 (20.7) | 42.0 (23.6)

ADVERSE EVENTS:
Time Frame: 6 months following surgery
Arm/Group | Bilateral GPi DBS Surgery Under General Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes